CLINICAL TRIAL: NCT06048731
Title: Enlighten Study: The EV-ICD Post Approval Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: PSR: EV-ICD PAS/PMCF
Record Dates: First submitted 2023-08-30; First posted 2023-09-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-02

CONDITIONS: Ventricular Arrhythmia; Tachycardia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Device: Defibrillation using EV-ICD — Device: Defibrillation using the Extravascular ICD (EV-ICD)

SUMMARY:
Medtronic is sponsoring Enlighten: The EV-ICD Post Approval Registry, to further confirm safety and effectiveness of EV-ICD in routine clinical practice, following commercial release of EV-ICD devices.

DETAILED DESCRIPTION:
The Enlighten Study is a global, prospective, observational, multi-site registry study. This study is conducted within Medtronic's post-market surveillance platform.

Eligibility for enrollment is based on market release dates for EV-ICD System within the geography in which the subject is enrolled.

Patients enrolled in the Enlighten Study will be prospectively followed for the life time of device post-implant or until registry closure, patient death or patient exit from the registry (i.e., withdrawal of consent).

Successfully implanted patients are expected to have scheduled follow-up visits per routine clinical care, at least annually, or as prompted by reportable adverse events. The total estimated registry duration is through lifetime of device.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient is intended to receive or be treated with a EV-ICD device System and must be enrolled prior to the EV-ICD device implant procedure

Exclusion Criteria:

* Patient who is, or is expected to be, inaccessible for follow-up
* Patient is excluded by local local law
* Patient is currently enrolled or plans to enroll in any concurrent drug and/or device study that may confound the PSR results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients intended to be implanted with a EV-ICD system are eligible for enrollment and all patients must be consented prior to implant. Geographies with regulatory approval for the EV-ICD system are eligible to enroll patients (see locations section). All patients enrolled and successfully implanted with an EV-ICD system will be followed for lifetime of device, unless a patient is exited from the registry due to an unavoidable reason such as death, physician discretion, or patient withdrawal of consent. If EV-ICD system is not successfully implanted, patients will be exited from the registry unless a EV-ICD System and/or implant procedure related event is identified, for which the patient will be followed until the event is resolved or no further actions need to be taken.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2037-10-31 (Estimated)

PRIMARY OUTCOMES:
Complication-free survival rate | 5 years
  To demonstrate 5-year Aurora EV-ICD major system-related complication-free survival > 79%

SECONDARY OUTCOMES:
System and/or procedure related complication-free survival | Procedure related complications assessed during and after the procedure/surgery; system related complications assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  To estimate the Aurora EV-ICD major system and/or procedure related complication-free survival probability as a function of time post-implant
Abnormal battery depletion complications | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Characterize the rate of abnormal battery depletion complications as a function of time post-implant
Summarize all device system revisions | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Summarize all device system revisions (e.g., reposition, replacement, explant) including reasons for modification and action taken
Patient deaths | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Summarize patient deaths
Patient demographics and baseline medical history | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Summarize patient demographics and baseline medical history
Characterize extracardiac pacing sensation | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Characterize extracardiac pacing sensation
Summarize ATP with spontaneous arrhythmias | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Summarize ATP with spontaneous arrhythmias
Characterize asystole pacing | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Characterize asystole pacing
Characterize sensing and detection | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Characterize sensing and detection
To characterize defibrillation shock effectiveness for terminating spontaneous VT/VF arrhythmia | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Characterize high voltage therapy effectiveness on device detected spontaneous ventricular episodes
Characterize lead location and lead motion at implant. | Assessed through the study completion (12 years average), and assessed every year (1 year, 2 years, 3 years, … 12 years)
  Characterize lead location and lead motion at implant.

CONTACTS AND LOCATIONS:
Locations (131):
- United States (57):
  - Cardiology Associates Medical Group, Huntington Park, California
  - Sequoia Hospital, Redwood City, California
  - University of California San Diego, San Diego, California
  - Stanford Hospital & Clinics, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Baptist Health, Jacksonville, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Wellstar Research Institute, Marietta, Georgia
  - Deaconess Specialty Physicians, Newburgh, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Norton Heart and Vascular Institute, Louisville, Kentucky
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Metropolitan Cardiology Consultants, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Health System, Kansas City, Missouri
  - University of Kansas Medical Center Research Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Virtua Health, Marlton, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Northwell Health South Shore University Hospital, Bay Shore, New York
  - Northwell Health Huntington Hospital, Huntington, New York
  - Northwell Health North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYU Langone Medical Center, New York, New York
  - New York-Presbyterian Hospital Columbia University, New York, New York
  - New York - Presbyterian Hospital / Weill Cornell Medical Center, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Northwell Health Staten Island University Hospital, Staten Island, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - The Christ Hospital Health Network CRD, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - OhioHealth Research Institute (OHRI), Columbus, Ohio
  - Saint Luke's University Health Network, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Shadyside, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Passavant, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - The Stern Cardiovascular Foundation, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Consultants in Cardiology (Fort Worth), Dallas, Texas
  - Heart Center of North Texas, Fort Worth, Texas
  - Baylor Research Institute, Plano, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Austria (4):
  - LKH - Universitätsklinikum Graz, Graz
  - Aö Landeskrankenhaus - Universitätskliniken Innsbruck, Innsbruck
  - Kepler Universitätsklinikum Med Campus III, Linz
  - Allgemeines Krankenhaus - Universitätskliniken Wien, Vienna
- Belgium (2):
  - AZ Sint Jan Brugge-Oostende av, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
- Canada (4):
  - University Of Calgary, Calgary, Alberta
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumo, Québec, Quebec
  - McGill University Health Centre (MUHC), Montreal
- Nemocnice Na Homolce, Prague, Czechia
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense
- Helsinki University Hospital, Helsinki, Finland
- France (11):
  - Centre Hospitalier Universitaire de Clermont-Ferrand - Gabriel-Montpied, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Grenoble - Site Nord, La Tronche
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - OC Santé - Clinique du Millénaire, Montpellier
  - Hôpital Guillaume et René Laënnec - CHU de Nantes, Nantes
  - Hopital Pitie-Salpetriere AP-HP, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHRU de Tours - Hôpital Trousseau, Saint-Avertin
- Germany (5):
  - Herz- und Diabeteszentrum NRW - Ruhr-Universität Bochum, Bad Oeynhausen
  - Elektrophysiologie Bremen - Im Klinikum Links der Weser, Bremen
  - Medizinische Hochschule Hannover, Hanover
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Eberhard Karls Universität Tübingen - Universitätsklinikum Tübingen, Tübingen
- Greece (2):
  - Hippokration General Hospital of Athens, Athens
  - George Papanikolaou General Hospital, Thessaloniki
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Semmelweis Egyetem AOK, Budapest, Hungary
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (5):
  - Azienda Ospedaliera - Universitaria Consorziale Policlinico di Bari, Bari
  - Policlinico Di Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliera Ospedale Niguarda Cà Granda, Milan
  - Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliera San Gerardo, Monza
- Chest Disease Hospital, Kuwait City, Kuwait
- Netherlands (7):
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - St Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
  - HagaZiekenhuis - Locatie Leyweg, The Hague
- Christ Church Hospital, Christchurch, New Zealand
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Narodowy Instytut Kardiologii - Stefana kardynała Wyszyńskiego, Warsaw
  - Slaskie Centrum Chorob Serca, Zabrze
- Portugal (2):
  - Centro Hospitalar de Lisboa Ocidental, E.P.E. Hospital de Santa Cruz, Carnaxide
  - Hospital de Santa Maria-Centro Hospitalar Lisboa Norte, EPE, Lisbon
- Saudi Arabia (2):
  - King Fahad Armed Forces Hospital, Jeddah
  - King Faisal Specialist Hospital & Research Centre, Riyadh
- Spain (7):
  - Hospital Universitario da Coruña, A Coruña
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario y Politécnico La Fe, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skånes Universitetssjukhus, Skåne
- Switzerland (5):
  - Universitätsspital Basel, Basel
  - Inselspital - Universitätsspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Istituto Cardiocentro Ticino, Lugano
  - UniversitätsSpital Zürich, Zurich
- United Kingdom (2):
  - Glenfield Hospital, Leicester
  - Kings College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boersma LVA, Amin A, Clementy N, Duncker D, Engel G, Epstein L, Kuriachan V, Frazier-Mills C, Gwechenberger M, Nishii N, Lande J, Wiggenhorn C, Crozier I. Design of a post-market registry for the extravascular implantable cardioverter-defibrillator: The Enlighten Study. Heart Rhythm O2. 2024 Oct 16;6(1):64-69. doi: 10.1016/j.hroo.2024.09.022. eCollection 2025 Jan. PMID 40224263